CLINICAL TRIAL: NCT02279342
Title: the Effect of Febuxostat on Coronary Plaque Volume in Patients With Chronic Stable Angina and Hyperuricemia
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Entry were insufficient as expected.
Sponsor: Yokohama City University Medical Center (Other)
Responsible Party: Principal Investigator, Kiyoshi Hibi, associate professor of medicine, Yokohama City University Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D1407027
Record Dates: First submitted 2014-08-14; First posted 2014-10-31 (Estimated); Last update posted 2017-08-03 (Actual); Status verified 2017-08

CONDITIONS: Coronary Artery Disease
Keywords: Coronary artery disease; hyperuricemia; coronary plaque volume; IVUS
MeSH Terms: conditions — Coronary Artery Disease; Hyperuricemia | interventions — Febuxostat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Non febuxostat treatment group (No Intervention): No febuxostat treatment
- Febuxostat treatment group (Experimental): once daily after breakfast
  Interventions: Drug: Febuxostat

INTERVENTIONS:
Drug: Febuxostat — The starting dose of the febuxostat will be 10mg /day. The dose will be increased to 20 mg/day at week 4 and finally titrated to 40 mg/day at week 8.
  Arms: Febuxostat treatment group

SUMMARY:
The purpose of this study is to investigate the effects of febuxostat on coronary plaque volume in patients with chronic stable angina and hyperuricemia.

DETAILED DESCRIPTION:
Patients with stable angina and hyperuricemia who undergo percutaneous coronary intervention (PCI) with intravascular ultrasound (IVUS) are enrolled. Participants will be randomly assigned to one of the two treatment groups.

Febuxostat group and A lifestyle modification group. At 8-12 months, routine follow up angiography and IVUS interrogation as well as endothelial function and several bio markers will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 20 years of age or older at enrollment who are able to visit
2. Patients with chronic stable angina who have severe coronary stenosis wich require PCI.
3. Patients who have at least one coronary plaque (≧ 500μm in thickness or % plaque of 20% or more) at the non-culprit vessels.
4. Patients with hyperuricemia, who have a serum uric acid level >7.0mg/dL within 2 months prior to enrollement.
5. Patients who personally given written informed consent to participate in this study.

Exclusion Criteria:

1. Patients who had undergone previous PCI for the lesion under investigation.
2. Patients with gouty tophus, or patients with subjective symptoms of gouty arthritis within 1 year prior to enrollment.
3. Patients with a previous history of hypersensitivity to febuxostat or allopurinol.
4. Patients with serious kidney disease, Acute kidney disease, nephrotic syndrome, dialysis patients, kidney transplant patients, eGFR < 30 mL/min/1.73m2, etc.
5. Patients with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) 2 or more times the upper limit of normal.
6. Patients on any of the following medications at enrollment Mercaptopurine hydrate, azathioprine, vidarabine, or didanosine.
7. Patients who receive any of the following medications for the treatment of hyperuricemia within 1 month prior to enrollment Allopurinol, benzbromarone, probenecid, bucolome, topiroxostat, or febuxostat.
8. Patients otherwise judged by the principal or sub-investigator to be unsuitable for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-10; Primary Completion 2017-03-31 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
The percent changes in coronary plaque volume obtained by IVUS from baseline to follow up | 8-12 months
The percent changes in integrated backscatter signal obtained by integrated backscatter IVUS from baseline to follow up | 8-12

SECONDARY OUTCOMES:
absolute changes of coronary plaque volume by IVUS from baseline to follow up | 8-12 months
absolute and percent changes in minimal lumen diameter and percent stenosis by QCA from baseline to follow up | 8-12 months
changes in plaque characteristics assessed by IVUS from baseline to follow up | 8-12 months
changes in serum uremic values and inflammatory markers from baseline to follow up | 8-12 months
prognosis(death, ACS, restenosis) | 8-12 months
nominal changes in plaque burden assessed by IVUS from baseline to follow up | 8-12 months
nominal changes in plaque burden adjusting for analyzed length assessed by IVUS from baseline to follow up | 8-12 months

CONTACTS AND LOCATIONS:
Overall Officials: Kiyoshi Hibi, MD, Study Chair — Yokohama City University Medical Center
Locations (1):
- Yokohama City University Medical Center, Yokohama, Kanagawa, Japan

IPD SHARING:
Plan to Share IPD: No